CLINICAL TRIAL: NCT01355276
Title: A Randomized, Double-blind, Double-dummy, Active Drug Parallel Controlled, Multi-center Clinical Trial on the Efficacy and Safety of Cinitapride Tablets in the Treatment of Mild to Moderate Functional Dyspepsia
Brief Title: Efficacy and Safety of Cinitapride Tablets in the Treatment of Mild to Moderate Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai China Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYWC100602
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Dyspepsia
Keywords: Cinitapride; efficacy; safety; mild to moderate functional dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — cinitapride; Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cinitapride
- 2 (Active Comparator)
  Interventions: Drug: domperidone

INTERVENTIONS:
Drug: Cinitapride — cinitapride 1 mg for each dose, 3 mg/daily, for 4 weeks
  Arms: 1
Drug: domperidone — 10 mg for each dose ,30 mg/daily, for 4 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to compare Cinitapride tablets with domperidone tablets (motilium), and to evaluate the efficacy and safety of Cinitapride tablets in the treatment of mild to moderate functional dyspepsia.

ELIGIBILITY:
Inclusion:

1. Aged between 18~65 years, both males and females;
2. Patients with symptoms of mild to moderate functional dyspepsia;
3. Symptoms related to dyspepsia were developed 6 months ago and early satiety or/and discomfort after meal were developed in the past 3 months;
4. Gastrointestinal malignancy, peptic ulcer, liver, gallbladder and pancreas diseases were excluded through gastroscopy, B-ultrasonography and laboratory examination within 4 weeks prior to administration (endoscopy results considered to be clinically unrelated will not be excluded, such as small hiatal hernia and chronic nonatrophic pangastritis);
5. Patient has signed informed consent form.

Exclusion criteria

1. Patients with gastroesophageal reflux and/or irritable bowel syndrome;
2. Acid regurgitation more than once per week;
3. Previously received abdominal surgery (except appendectomy and herniorrhaphy);
4. A history of gastric or duodenal ulcer;
5. Patients with depression and anxiety neurosis;
6. Patients with arrhythmia;
7. QTc more than 0.5s;
8. Hepatic and renal insufficiency: AST or/and ALT equal to or above 1.5 times of the upper normal limit; Cr above the upper normal limit;
9. Pathological lactorrhea;
10. Patients with alcohol abuse (daily alcohol intake more than 40g), drug dependence or neuropsychiatric disorders that are difficult to control, as well as others who are not appropriate to participate in a drug trial;
11. Pregnant or lactating women;
12. Patients who require other therapy to change gastrointestinal mobility;
13. Patients who are participating or participated in other drug clinical trial within 3 months prior to entry;
14. Known to be allergic to cinitapride; Patients who are considered by investigators to be inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response rate of overall symptom improvement after 4-weeks treatment | 4 weeks

SECONDARY OUTCOMES:
Percentage change of overall symptom score of functional dyspepsia from baseline after 2 and 4 weeks treatment | 2 and 4 weeks
Response rate after 2 weeks treatment | 2 weeks
Percentage change of individual symptom score (early satiety, discomfort with fullness after meal, flatulence, epigastric pain, epigastric burning, nausea, vomiting and belching) after 2 and 4 weeks treatment compared with the baseline | 2 and 4 weeks
Changes of gastric emptying in some patients after 4-week treatment | 4 weeks
Patient's global subjective assessment (Likert scale score) after 2 and 4 weeks treatment | 2 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Principal Investigator — Changhai Hospital
Locations (13):
- China (13):
  - The First Affiliated Hospital of Anhui medical university, Hefei, Anhui
  - Huazhong University of Science and Technology of Tongji Hospital Affiliated Tongji Medical School, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Changzhou First People?s Hospital, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Changhai Hospital, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - The Second Affiliated Hospital of Suzhou University, Suzhou
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Tianjin Medical University General Hospital, Tianjin

REFERENCES:
- [Derived] Du Y, Su T, Song X, Gao J, Zou D, Zuo C, Xie W, Wang B, Zhang Z, Xu J, Tian D, Luo H, Zhang Z, Wang S, Chen J, Guo J, Gong L, Ding Y, Li Z. Efficacy and safety of cinitapride in the treatment of mild to moderate postprandial distress syndrome-predominant functional dyspepsia. J Clin Gastroenterol. 2014 Apr;48(4):328-35. doi: 10.1097/MCG.0000000000000033. PMID 24440931